CLINICAL TRIAL: NCT01025843
Title: A Single Dose Study to Evaluate the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of MK5478 in Subjects and in Patients With Hypertension
Brief Title: Safety and Tolerability of MK-5478 in Participants With Hypertension (5478-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5478-001; 2009-016048-38 (EudraCT Number)
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Pbo → 5 mg → Candesartan → 24 mg → 38 mg (Experimental): Placebo in Period 1; 5 mg MK-5478 in Period 2; Candesartan in Period 3; 24 mg MK-5478 in Period 4; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- 1 mg → 5 mg → 12 mg → Candesartan → Pbo (Experimental): 1 mg MK-5478 in Period 1; 5 mg MK-5478 in Period 2; 12 mg MK-5478 in Period 3; Candesartan in Period 4; and Placebo in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- 1 mg → Candesartan → Pbo → 24 mg → 38 mg (Experimental): 1 mg MK-5478 in Period 1; Candesartan in Period 2: Placebo in Period 3; 24 mg MK-5478 in Period 4; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- 1 mg → 5 mg → 12 mg → Pbo → Candesartan (Experimental): 1 mg MK-5478 in Period 1; 5 mg MK-5478 in Period 2; 12 mg MK-5478 in Period 3; Placebo in Period 4; and Candesartan in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- Pbo→ 8 mg→ 18 mg → 2 mg fed→Candesartan (Experimental): Placebo in Period 1; 8 mg MK-5478 in Period 2; 18 mg MK-5478 in Period 3; 2 mg MK-5478 in Period 4 with a high fat meal; and Candesartan in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- 2 mg→Pbo → Candesartan → Pbo fed→38 mg (Experimental): 2 mg MK-5478 in Period 1; Placebo in Period 2; Candesartan in Period 3; Placebo in Period 4 with a high fat meal; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- 2 mg→Candesartan→Pbo→Candesartan fed→38 mg (Experimental): 2 mg MK-5478 in Period 1; Candesartan in Period 2; Placebo in Period 3; Candesartan in Period 4 with a high fat meal; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- 2 mg → 8 mg → 18 mg → 2 mg fed → Pbo (Experimental): 2 mg MK-5478 in Period 1; 8 mg MK-5478 in Period 2; 18 mg MK-5478 in Period 3; 2 mg MK-5478 in Period 4 with a high fat meal; and Placebo in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- Candesartan→8 mg→ 18 mg →2 mg fed→38 mg (Experimental): Candesartan in Period 1; 8 mg MK-5478 in Period 2; 18 mg MK-5478 in Period 3; 2 mg MK-5478 in Period 4 with a high fat meal; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo
- Candesartan→Pbo → 12 mg → 24 mg→38 mg (Experimental): Candesartan in Period 1; Placebo in Period 2; 12 mg MK-5478 in Period 3; 24 mg MK-5478 in Period 4; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
  Interventions: Drug: MK-5478; Drug: Comparator: Candesartan cilexetil; Drug: Comparator: Pbo

INTERVENTIONS:
Drug: MK-5478 — In Part I: Single dose administration of MK-5478 oral capsules, total doses of 1, 2, 5, 8, 12, 18, 24 or 38 mg.
Drug: Comparator: Candesartan cilexetil — Single dose administration of candesartan, 32 mg oral tablet
  Other Names: Atacand/Amias
Drug: Comparator: Pbo — Placebo

SUMMARY:
This is a two part introductory clinical trial with MK-5478. Part I will evaluate the safety, tolerability and pharmacokinetics and pharmacodynamics of MK-5478 in young, healthy males. Part II will evaluate the safety, tolerability and pharmacodynamic effects of MK-5478 in participants with hypertension. The primary hypothesis is that single oral doses of MK-5478 are sufficiently safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

Part I:

* Is a male between 18 to 50 years of age
* Is in good health
* Is a non-smoker

Part II:

* Is male of non-child bearing potential between 18 and 50 years of age
* Has hypertension (high blood pressure)

Exclusion Criteria:

Part I and Part II:

* Has a history of stroke, seizures or major neurological disorder
* Has a history of cancer
* Has a history of any cardiovascular disease
* Is unable to refrain from the use of any prescription or non-prescription drugs
* Consumes excessive amounts of alcohol or caffeine
* Has had major surgery, donated blood or participated in another investigational study in the past 4 weeks

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2010-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=5478-001&kw=5478-001&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Part II of this study was planned. However, since the efficacy criteria for advancing to Part II were not met in Part I, this study was considered completed with the completion of Part I. Therefore participants were not recruited for Part II.
Groups:
- 1 mg → Candesartan → Pbo → 24 mg → 38 mg: 1 mg MK-5478 in Period 1; Candesartan in Period 2: Placebo in Period 3; 24 mg MK- 5478 in Period 4; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
- Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan: Placebo in Period 1; 8 mg MK-5478 in Period 2; 18 mg MK-5478 in Period 3; 2 mg MK-5478 in Period 4 with a high fat meal; and Candesartan in Period 5. There was a minimum 7 days washout between periods.
- 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg: 2 mg MK-5478 in Period 1; Placebo in Period 2; Candesartan in Period 3; Placebo in Period 4 with a high fat meal; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
- 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg: 2 mg MK-5478 in Period 1; Candesartan in Period 2; Placebo in Period 3; Candesartan in Period 4 with a high fat meal; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
- Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg: Candesartan in Period 1; 8 mg MK-5478 in Period 2; 18 mg MK-5478 in Period 3; 2 mg MK-5478 in Period 4 with a high fat meal; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods.
- Candesartan → Pbo → 12 mg → 24 mg → 38 mg: Candesartan in Period 1; Placebo in Period 2; 12 mg MK-5478 in Period 3; 24 mg MK- 5478 in Period 4; and 38 mg MK-5478 in Period 5. There was a minimum 7 days washout between periods
Period: Period 1
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 1
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 2
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 3
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout 4
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg
Started | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Pbo → 5 mg → Candesartan → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Candesartan → Pbo | 1 mg → Candesartan → Pbo → 24 mg → 38 mg | 1 mg → 5 mg → 12 mg → Pbo → Candesartan | Pbo → 8 mg→ 18 mg → 2 mg Fed → Candesartan | 2 mg→Pbo → Candesartan → Pbo Fed → 38 mg | 2 mg→Candesartan→ Pbo → Candesartan Fed → 38 mg | 2 mg → 8 mg → 18 mg → 2 mg Fed → Pbo | Candesartan→8 mg→ 18 mg → 2 mg Fed → 38 mg | Candesartan → Pbo → 12 mg → 24 mg → 38 mg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 20
Age, Continuous [Median (Full Range); unit: Years] | 46.5 [46 to 47] | 38.5 [29 to 48] | 46.0 [45 to 47] | 35.0 [21 to 49] | 37.5 [36 to 39] | 44.5 [40 to 49] | 48.0 [46 to 50] | 46.5 [44 to 49] | 45.0 [42 to 48] | 39.0 [38 to 40] | 45.5 [21 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Adverse Events (AEs)
Description: An AE is any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, is also an AE.
Time Frame: Up to 14 days after administration of last dose of study drug (up to Day 52)
Population: All participants who received at least one dose of the investigational drug, according to the treatment(s) they actually received; according to study drug taken at time of the event and not by randomly assigned sequence.
Measure: Number; unit: Participants
Groups:
- MK-5478 1 mg: A single dose of 1 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 2 mg: A single dose of 2 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 5 mg: A single dose of 5 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 8 mg: .A single dose of 8 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 12 mg: A single dose of 12 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 18 mg: A single dose of 18 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 24 mg: A single dose of 24 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 38 mg: A single dose of 38 mg MK-5478 in capsule form was orally administered during a treatment period
- MK-5478 2 mg - Fed: A single dose of 2 mg MK-5478 in capsule form was orally administered during a treatment period, preceded by a high fat breakfast
- Candesartan 32 mg: A single dose of 32 mg Candesartan in tablet form was orally administered during a treatment period
- Candesartan 32 mg - Fed: A single dose of 32 mg Candesartan in tablet form was orally administered during a treatment period, preceded by a high fat breakfast
- Candesartan Placebo: A single dose of Candesartan placebo in tablet form was orally administered during a treatment period
- MK-5478 Placebo: A single dose of MK-5478 Placebo in capsule form was orally administered during a treatment period
Arm/Group | MK-5478 1 mg | MK-5478 2 mg | MK-5478 5 mg | MK-5478 8 mg | MK-5478 12 mg | MK-5478 18 mg | MK-5478 24 mg | MK-5478 38 mg | MK-5478 2 mg - Fed | Candesartan 32 mg | Candesartan 32 mg - Fed | Candesartan Placebo | MK-5478 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 15 | 2 | 2 | 16
Participants | 5 | 3 | 3 | 4 | 4 | 3 | 2 | 2 | 1 | 9 | 0 | 1 | 6

2. Primary Outcome: Number of Participants Who Discontinued Treatment Due to an AE
Description: as for outcome 1
Time Frame: Up to 24 hours after administration of study drug
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | MK-5478 1 mg | MK-5478 2 mg | MK-5478 5 mg | MK-5478 8 mg | MK-5478 12 mg | MK-5478 18 mg | MK-5478 24 mg | MK-5478 38 mg | MK-5478 2 mg - Fed | Candesartan 32 mg | Candesartan 32 mg - Fed | Candesartan Placebo | MK-5478 Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 15 | 2 | 2 | 16
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC 0-infinity) of MK-5478 and Candesartan
Description: Blood was collected at the following time points: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, and 48 hours post-dose in order to measure AUC 0-infinity of MK-5478 and Candesartan
Time Frame: Pre-dose and up to 48 hours postdose
Population: In order to keep the study blinded, the scheduled number of treated participants rather than the actual number of treated participants were analyzed; according to the scheduled study drug and not by randomly assigned sequence.
Measure: Mean (Standard Deviation); unit: umol.hr/L
Arm/Group | MK-5478 1 mg | MK-5478 2 mg | MK-5478 5 mg | MK-5478 8 mg | MK-5478 12 mg | MK-5478 18 mg | MK-5478 24 mg | MK-5478 38 mg | MK-5478 2 mg - Fed | Candesartan 32 mg | Candesartan 32 mg - Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 2
umol.hr/L | 0.236 (0.141) | 0.494 (0.202) | 1.87 (0.538) | 1.80 (0.436) | 1.36 (0.448) | 2.23 (0.582) | 3.15 (1.55) | 4.50 (0.857) | 0.504 (0.07) | 5.89 (1.38) | 4.46 (0.314)

4. Secondary Outcome: Change From Baseline in Aortic Augmentation Index (AIx) of MK-5478 and Candesartan
Description: Central blood pressure (CBP) parameters will be measured and used to derive the aortic augmentation index (AIx). The AIx quantifies the contribution of back-reflected outgoing systolic pressure waves to late-systolic central blood pressure, which increases with decreasing aortic compliance. AIx is measured by pulse wave analysis using the SphygmoCor System supplied by AtCor Medical. Results with a > 5% decrease in AIx were planned for analysis; results with a < 5% decrease in AIx were not analysed.
Time Frame: Baseline and 1 to 3 hours postdose
Population: Results were not analyzed because none showed a > 5% decrease in AIx.
Arm/Group | MK-5478 1 mg | MK-5478 2 mg | MK-5478 5 mg | MK-5478 8 mg | MK-5478 12 mg | MK-5478 18 mg | MK-5478 24 mg | MK-5478 38 mg | MK-5478 2 mg - Fed | Candesartan 32 mg | Candesartan 32 mg - Fed
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-5478 and Candesartan
Description: Blood was collected at the following time points: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 36, and 48 hours post-dose in order to measure the Cmax of MK-5478 and Candesartan
Time Frame: Pre-dose and up to 48 hours postdose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | MK-5478 1 mg | MK-5478 2 mg | MK-5478 5 mg | MK-5478 8 mg | MK-5478 12 mg | MK-5478 18 mg | MK-5478 24 mg | MK-5478 38 mg | MK-5478 2 mg - Fed | Candesartan 32 mg | Candesartan 32 mg - Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 16 | 2
µmol/L | 0.0291 (0.012) | 0.0573 (0.0206) | 0.254 (0.0588) | 0.227 (0.0630) | 0.120 (0.0332) | 0.245 (0.0634) | 0.321 (0.206) | 0.532 (0.154) | 0.0553 (0.00891) | 0.476 (0.194) | 0.451 (0.0641)

ADVERSE EVENTS:
Time Frame: 14 days after administration of last dose of study drug (up to Day 52)
Description: All participants who received at least one dose of the investigational drug, according to the treatment(s) they actually received; according to study drug taken at time of the event and not by randomly assigned sequence.
Arm/Group | MK-5478 1 mg | MK-5478 2 mg | MK-5478 5 mg | MK-5478 8 mg | MK-5478 12 mg | MK-5478 18 mg | MK-5478 24 mg | MK-5478 38 mg | MK-5478 2 mg - Fed | MK-5478 Placebo | Candesartan 32 mg | Candesartan 32 mg - Fed | Candesartan Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/16 | 0/15 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 3/6 | 4/6 | 4/6 | 3/6 | 2/6 | 2/5 | 1/6 | 6/16 | 9/15 | 0/2 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-5478 1 mg (N=6) | MK-5478 2 mg (N=6) | MK-5478 5 mg (N=6) | MK-5478 8 mg (N=6) | MK-5478 12 mg (N=6) | MK-5478 18 mg (N=6) | MK-5478 24 mg (N=6) | MK-5478 38 mg (N=5) | MK-5478 2 mg - Fed (N=6) | MK-5478 Placebo (N=16) | Candesartan 32 mg (N=15) | Candesartan 32 mg - Fed (N=2) | Candesartan Placebo (N=2)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loose stools (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts,or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.